CLINICAL TRIAL: NCT03697057
Title: Computerised 4-choice Reaction Time Test for the Measurement of Psychomotor Recovery After General Anaesthesia
Brief Title: 4-choice Reaction Time Test for the Measurement of Psychomotor Recovery After General Anaesthesia
Acronym: 4CRT_Ane
Status: Completed | Type: Observational
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Other Study IDs: III UV 03/05
Record Dates: First submitted 2018-10-01; First posted 2018-10-05 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Postoperative Complications
Keywords: postoperative recovery; psychomotor function; measurement
MeSH Terms: conditions — Postoperative Complications | interventions — Anesthesia, General

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients: Patients scheduled for elective ambulatory gynaecological surgery, which was performed under standardised general anaesthesia
  Interventions: Procedure: General anaesthesia
- healthy volunteers: Female healthy volunteers matched to the patient group regarding the age

INTERVENTIONS:
Procedure: General anaesthesia — Standard general anaesthesia for gynecologic surgery in patient group
  Groups: patients

SUMMARY:
The recovery of patients after general anaesthesia is usually estimated by using clinical signs and scores. Since there is a lack of the agreed objective methods for assessing cognitive and psychomotor recovery after general anaesthesia in ambulatory settings, the aim of this study was to evaluate three psychological tests for this purpose. Patients, who were scheduled for ambulatory gynaecological surgery, underwent 3 standard psychological tests before (T1), 15 minutes after the surgery (T2) and on discharge from the recovery room (T3). The tests used were Wechsler memory scale (test 1, working memory capacity), d2 - test (test 2, concentration endurance) and computer-based 4-choice-reaction time (4CRT, test 3, reaction time) as well as Postanesthesia Discharge Scoring System (PADSS). The same test battery was used in healthy female volunteers, all test results were compared at the different time points.

ELIGIBILITY:
Inclusion Criteria:

* consecutive patients scheduled for ambulatory gynaecologic surgery
* age of 18 to 60 years
* a physical status I-II according to American Society of Anesthesiologists (ASA) classification
* fluency in German language and the ability to perform all tests

Exclusion Criteria:

* chronic consume of analgesics, psychotropic drugs, sedatives or alcohol
* if the ambulatory surgery lasted more than 60 minutes
* if the schema of standardised general anaesthesia was changed
* if the ambulatory setting was changed and the patients unexpectedly remained over night in the hospital.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Consecutive patients scheduled for ambulatory gynaecologic surgery were asked to participate in the study during the routine informed consent process for anaesthesia. The inclusion criteria are listed in previous Section. A group of healthy female volunteers, meeting the eligibility criteria, completed the same study procedure without a surgery at three matched time points; none of them was taking any medication at the time of the study. Written informed consent was obtained from all individuals.
Sampling Method: Non-Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2008-03 (Actual); Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
4CRT_15_min | 15 minutes after the end of surgery
  Change of four choice reaction time (4CRT) at 15 minutes after surgery from baseline

SECONDARY OUTCOMES:
PADSS (Patient Discharge Scoring System) | Measured 60 minutes after the end of surgery
  Post Anaesthetic Discharge Scoring System (PADSS) is a clinically-based, objective scoring system used to measure the home readiness of patients following day surgery. PADSS consists of six criteria: ambulation, circulation (blood pressure monitoring), nausea/vomiting, pain and surgical bleeding bleeding. Each criterion is given a score ranging from 0 to 2, maximal score is 10. Only patients who achieve a score of 9 or more are considered ready for discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hesse, MD, Principal Investigator — University Medicine of Greifswald
Locations (1):
- University Medicine of Greifswald, Greifswald, Germany

IPD SHARING:
Plan to Share IPD: No
We will send the IPD on request via email.